CLINICAL TRIAL: NCT07224672
Title: A Phase 2, Open-label, Single-arm, Proof-of-concept Study Evaluating the Efficacy and Safety of Belantamab Mafodotin Administered in Combination With Cyclophosphamide, Bortezomib, and Dexamethasone in Adult Participants With Newly Diagnosed Amyloid Light Chain Amyloidosis (ALANIS)
Brief Title: A Study to Evaluate the Efficacy and Safety of Belantamab Mafodotin in Combination With Cyclophosphamide, Bortezomib, and Dexamethasone in Adult Participants With Newly Diagnosed Amyloid Light Chain (AL) Amyloidosis
Acronym: ALANIS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 223963; 2025-522803-60 (Other: EU CT Number)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2025-10-31; First posted 2025-11-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Amyloidosis
Keywords: Amyloid light chain amyloidosis; Bortezomib; Cyclophosphamide; Dexamethasone; Proof of concept study
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — belantamab mafodotin; Cyclophosphamide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab mafodotin + cyclophosphamide, bortezomib, and dexamethasone (CyBorD) (Experimental): Adult participants with newly diagnosed amyloid light chain (AL) amyloidosis will receive Belantamab mafodotin in combination with CyBorD.
  Interventions: Drug: Belantamab mafodotin; Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered
Drug: Cyclophosphamide — Cyclophosphamide will be administered
Drug: Bortezomib — Bortezomib will be administered
Drug: Dexamethasone — Dexamethasone will be administered

SUMMARY:
The study aims to evaluate the efficacy and safety of belantamab mafodotin in combination with cyclophosphamide, bortezomib, and dexamethasone in adult participants with newly diagnosed (ND) AL amyloidosis .

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years of age or the legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the informed consent form (ICF).
* Has histologically confirmed newly diagnosed primary AL amyloidosis according to the following criteria:

  * Presence of an amyloid-related systemic syndrome with 1 or more organs involved (e.g., renal, liver, heart, gastrointestinal tract, or peripheral nerve involvement, as per consensus guidelines).
  * Positive amyloid staining by Congo red stain with apple green birefringence on polarized light microscopy in any tissue (e.g., fat aspirate, bone marrow [BM], or organ biopsy), AND Characteristic appearance by electron microscopy and confirmatory immunohistochemistry or AL amyloidosis typing by mass spectrometric proteomic analysis of the amyloid deposits or amyloid-typing by immunofluorescence
  * Evidence of a monoclonal plasma cell proliferative disorder (serum or urine monoclonal protein, abnormal free light chain [FLC] ratio, or clonal plasma cells in the BM)
* Measurable clonal disease as defined by at least 1 of the following:

  * Serum monoclonal protein >=0.5 grams per deciliter (g/dL) by protein electrophoresis (routine serum protein electrophoresis and immunofixation performed at central laboratory),
  * Serum FLC >=5.0 milligram per deciliter (mg/dL) with an abnormal kappa:lambda ratio or the difference between involved and difference between amyloidogenic (involved) and non-amyloidogenic (uninvolved) FLC concentrations (dFLC) >=5 mg/dL.
* Not considered candidate for high-dose chemotherapy with autologous stem cell transplantation (ASCT) as part of first line of therapy, as per consensus guidelines
* Is willing to use adequate contraception. Contraceptive use by male and female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Is capable of giving signed informed consent
* Has an Eastern Cooperative Oncology Group performance status of 0, 1 or 2, with no deterioration in the 2 weeks before enrollment.
* Has adequate hematologic, hepatic and renal function as per the protocol

Exclusion Criteria:

* Has a previous or current diagnosis of plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes (POEMS) syndrome or symptomatic multiple myeloma (MM), as per International Myeloma Working Group criteria for MM including the presence of lytic bone disease (>=1 osteolytic lesion on imaging tests skeletal radiography, Computed Tomography [CT] scan, positron emission tomography/CT scan or Magnetic resonance imaging [MRI]), plasmacytomas, or clonal BM plasma cells >=60%. Note: A participant with a serum FLC ratio ≥100 or <0.01 who otherwise does not fulfil criteria for MM will be eligible.
* Has Immunoglobulin M (IgM)-related AL amyloidosis.
* Has any form of non-AL amyloidosis, including wild type or mutated (Transthyretin amyloidosis [ATTR]) amyloidosis.
* Has evidence of significant cardiovascular (CV) conditions as specified below:

  * New York Heart Association (NYHA) classification IIIb or IV heart failure.
  * Heart failure that in the opinion of the investigator is caused by ischemic heart disease (e.g., prior myocardial infarction with documented history of cardiac enzyme elevation and electrocardiogram [ECG] changes) or uncorrected valvular disease and not primarily due to AL amyloidosis cardiomyopathy.
  * In-participant admission to a hospital for unstable angina or myocardial infarction within the last 3 months prior to screening or percutaneous cardiac intervention with recent stent within last 3 months prior to screening or coronary artery bypass grafting within the last 3 months prior to screening
  * Participants with current evidence of clinically significant untreated arrhythmia(s), including clinically significant ECG abnormalities including second-degree (Mobitz Type II) or third-degree atrioventricular block.
  * Participants with a history of sustained ventricular tachycardia or aborted ventricular fibrillation or with a history of atrioventricular nodal or sinoatrial nodal dysfunction for which a pacemaker/implantable cardioverter-defibrillator is indicated but not placed (participants who do have a pacemaker/implantable cardioverter-defibrillator are allowed on the study).
  * Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >450 millisecond (msec) or >480 msec for participants with bundle branch block. Participants who have a pacemaker may be included regardless of calculated QTc interval.
  * Supine systolic blood pressure <90 millimeters of mercury (mmHg), or symptomatic orthostatic hypotension, defined as a decrease in systolic blood pressure upon standing of >20 mmHg despite medical management (e.g., midodrine, fludrocortisones) in the absence of volume depletion.
  * Uncontrolled hypertension.
* Has Mayo stage 3B disease
* Has a current corneal epithelial disease except for mild punctate keratopathy.
* Has previous or concurrent malignancies other than AL amyloidosis, except for any other malignancy that has been considered medically stable for at least 2 years, after discussion with GSK medical monitor. The participant must not be receiving active therapy, other than hormonal therapy for this disease.
* Has major surgery within 2 weeks prior to the first dose of study interventions or has not recovered fully from surgery.
* Has any history of prior allogenic or autologous BM transplant or other solid organ transplant.
* Has known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to belantamab mafodotin, cyclophosphamide, bortezomib, boron or mannitol or any other components or excipients or other allergy that, in the opinion of the investigator or GSK medical monitor, contraindicates participation in the study.
* Has any serious and/or unstable medical or psychiatric disorder or other condition(s) (including laboratory assessment abnormalities) that could interfere with the participant's safety, obtaining of informed consent, or compliance with the study procedures.
* Has active infection or active bleeding.
* Has intolerance or contraindications to antiviral prophylaxis.
* Has known Human immunodeficiency virus (HIV) infection, unless the participant can meet all of the following criteria:

  * Established anti-retroviral therapy (ART) for at least 4 weeks and HIV viral load <400 copies/milliliter (mL) within the screening period.
  * Cluster of differentiation 4 plus (CD4+) T-cell (CD4+) counts >=350 cells/microliter.
  * No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the last 12 months.
* Has prior therapy for AL amyloidosis or MM, with the exception of 160 milligram (mg) dexamethasone (or equivalent corticosteroid) maximum exposure prior to enrollment.
* Has received any live or live-attenuated vaccine within 30 days prior to first dose of belantamab mafodotin
* Is currently enrolled or has participated in any other clinical study involving an investigational study intervention or any other type of interventional medical research within 28 days before enrollment.
* Has an alanine aminotransferase (ALT) value >2.5*upper limit of normal (ULN) or >3*ULN if hepatic involvement of AL amyloidosis
* Has a total bilirubin value >1.5*ULN
* Has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice
* Has documented presence of Hepatitis B surface antigen (HBsAg) and/or Hepatitis B core antibody (HBcAb) at screening or within 3 months prior to the first dose of study intervention.
* Has a positive hepatitis C antibody test result or positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention unless the participant can meet the following criteria:

  * RNA test negative.
  * Successful antiviral treatment (usually 8 weeks duration) is required, followed by a negative Hepatitis C virus RNA test after a washout period of at least 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-11 (Estimated); Primary Completion 2027-08-10 (Estimated); Study Completion 2032-02-04 (Estimated)

PRIMARY OUTCOMES:
Overall complete hematologic response (CHR) rate | Up to approximately 24 months
  The overall CHR rate is defined as the proportion of participants who achieve a CHR during or after study treatment initiation, as assessed by the investigator, according to the consensus guidelines for AL amyloidosis.

SECONDARY OUTCOMES:
Number of participants with non-serious adverse events and serious adverse events | Up to approximately 24 months
Number of participants with clinically significant changes in hematology, and chemistry parameters | Up to approximately 24 months
Number of participants with ocular findings on ophthalmic examination | Up to approximately 24 months
Organ response rate (OrRR) | Up to approximately 5 years
  OrRR is defined as the proportions of participants who achieve confirmed organ response (cardiac, renal, or liver) in each organ as per consensus guidelines.
Duration of CHR | Up to approximately 5 years
  Duration of CHR is defined for participants with CHR as the time from the date of initial documentation of CHR to the date of first documented evidence of hematologic progressive disease.
Maximum plasma concentration (Cmax) of belantamab mafodotin | Up to 24 months
Area under the concentration-time curve (AUC) of belantamab mafodotin | Up to 24 months
Cmax of Cysteine maleimidocaproyl monomethyl auristatin F (cys-mcMMAF) | Up to 24 months
AUC of cys-mcMMAF | Up to 24 months
Number of participants with positive anti-drug antibodies (ADAs) against belantamab mafodotin | Up to approximately 24 months
Titers of ADAs against belantamab mafodotin | Up to approximately 24 months
Major organ deterioration - progression-free survival (MOD-PFS) | Up to approximately 5 years
  MOD-PFS is defined as duration from the date of study treatment initiation to either hematologic progression, or renal or cardiac failure or death, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No